CLINICAL TRIAL: NCT04860193
Title: Audiovestibular Functions in Covid 19 Patients in Sohag Governate
Brief Title: Audio Vestibular Functions in COVID 19 Patients in Sohag Governate
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Yasmeen Ali Mohamed, Principal investigator, Sohag University
Other Study IDs: Soh-Med-21-04-14
Record Dates: First submitted 2021-04-18; First posted 2021-04-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is evidence that up to 30% of COVID-19 patients was reported with neurological manifestations such as impaired consciousness, headache, and dizziness have been reported in COVID-19 patients in addition, olfactory and taste alterations are common symptoms in patients affected by COVID-19.This study will be conducted to evaluate the effect of the novel coronavirus on audio-vestibular functions in confirmed COVID19 patients.

ELIGIBILITY:
Inclusion Criteria:

- Well educated patients Age: range between 20 to 50 years No previous history of hearing loss or otoneurologic disease

Well confirmed COVID 19 patients:

patients who were diagnosed with coronavirus from

* symptoms: fever, cough, generalized malaise, dyspnea.
* Laboratory finding: abnormalities have been observed in Complete blood count (CBC), high C-reactive protein and ferritin, elevated D-dimer.
* Imaging: Chest CT scan: bilateral ground glass opacities, crazy paving, and consolidation.
* nasopharyngeal swab for SARS-CoV-2 polymerase chain reaction testing (RT-PCR).

Exclusion Criteria:

* previous history of hearing loss or otoneurological disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The present study will include 100 of randomly selected patients who were had been confirmed to be infection with COVID 19 virus, age ranged from 20-50 years. The investigation will be done three months after infection and after being sure that the patient become noninfectious.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2023-03-18 (Actual)

PRIMARY OUTCOMES:
Basic audiological evaluation: | 3 months after infection
  Pure-tone audiometry.
Basic audiological evaluation: | 3 months after infection
  Acoustic immittance testing
Basic audiological evaluation: | 3 months after infection
  Speech audiometry
Auditory evoked potentials: | 3 months after infection
  Auditory brainstem response.
Auditory evoked potentials | 3 months after infection
  P300
Effect on vestibular functions | 3 months after infection
  Videonystagmography
Effect on vestibular functions | 3 months after infection
  Video Head Implus test VHIT.
Effect on vestibular functions | 3 months after infection
  Vestibular evoked myogenic potential.
Effect on vestibular functions | 3 months after infection
  Computerized Dynamic Posturography (CDP)

SECONDARY OUTCOMES:
Effect on cognitive functions | 3 months after infection
  Cognitive function assessment:
  By Montreal test
Vestibular questionnaire | 3 months after infection
  Dizziness Handicap Inventory (DHI).

CONTACTS AND LOCATIONS:
Overall Officials: Yasmeen Mohamed, Principal Investigator
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided